CLINICAL TRIAL: NCT02158182
Title: Comparison of Three Different Schemes:Lactulose, L-ornithine L-aspartate, or Rifaximin, Versus Placebo, as Primary Prophylaxis of the Development of Hepatic Encephalopathy After Acute Variceal Bleeding in Cirrhotic Patients
Brief Title: Lactulose, L-ornithine L-aspartate, or Rifaximin Versus Placebo for Preventing Hepatic Encephalopathy in Variceal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, MARIA DE FATIMA HIGUERA DE LA TIJERA, MD, MSc., Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DI/14/107/03/028
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy; Acute Variceal Bleeding; Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Lactulose; ornithylaspartate; Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- lactulose (Experimental)
  Interventions: Drug: Lactulose
- L-ornithine L-aspartate (Experimental)
  Interventions: Drug: L-ornithine L-aspartate
- Rifaximin (Experimental)
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactulose — 30 ml by mouth three times daily until melena resolved, then adjusted to dose-response to obtain two to three soft stools. Duration of therapy: 7 days
  Arms: lactulose
Drug: L-ornithine L-aspartate — 10 grams by intravenous way for 24 hours. Duration of therapy: 7 days
  Arms: L-ornithine L-aspartate
Drug: Rifaximin — 2 tablets (400mg) three times daily. Duration of therapy: 7 days
  Arms: Rifaximin
Drug: Placebo — Placebo (for lactulose) 30ml of dextrose solution by mouth three times daily, for 7 days.
  Placebo (for L-ornithine L-aspartate) saline solution 500ml by intravenous way for 24 hours, for 7 days.
  Placebo (for rifaximin) 2 dextrose tablets three times daily for 7 days.
  Arms: Placebo

SUMMARY:
The aim of this study is to determine whether lactulose, L-ornithine L-aspartate, and rifaximin are effective in the prevention of the development of hepatic encephalopathy in cirrhotic patients with acute variceal bleeding

ELIGIBILITY:
Inclusion Criteria:

-Cirrhotic patients with acute variceal bleeding, without minimal or clinical hepatic encephalopathy according to PHES, CFF and West-Haven criteria

Exclusion Criteria:

* Age under 18 year-old or over 65 year-old, with any other neuropsychiatric disorder or dementia, presence of active bacterial or fungal infections, receiving antibiotics for any cause, previous diagnosis of hepatic encephalopathy and receiving therapy with lactulose, rifaximin, L-ornithine L-aspartate, source of bleeding different from variceal origin, serum creatinine greater than 2.0 mg/dl or with chronic renal failure. Therapy in the previous six months with any of the drugs that will be used in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Development of clinical hepatic encephalopathy | 7 days
  Determined by West-Haven Criteria

SECONDARY OUTCOMES:
Development of minimal hepatic encephalopathy | 7 days
  Determined by psychometric hepatic encephalopathy score (PHES) and critical flicker frequency (CFF)

OTHER OUTCOMES:
Development of adverse effects | 7 days
  Side or adverse effect will be defined as an undesirable secondary effect which occurs in addition to the desired therapeutic effect of a drug or medication.
  Non serious side effect will be defined as an undesirable secondary effect that does not represents a risk for patient´s life or function.
  Particularly we will addressed: Diarrhea, bloating, nausea, vomiting, elevation of serum creatinine, flatulence, abdominal pain, constipation, headache, dizziness
  Serious side effect will be defined as an undesirable secondary effect that represents a risk for patient´s life or function.
  Particularly we will addressed: allergic reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Mexico, Mexico City, Mexico

REFERENCES:
- [Derived] Higuera-de-la-Tijera F, Servin-Caamano AI, Salas-Gordillo F, Perez-Hernandez JL, Abdo-Francis JM, Camacho-Aguilera J, Alla SN, Jimenez-Ponce F. Primary Prophylaxis to Prevent the Development of Hepatic Encephalopathy in Cirrhotic Patients with Acute Variceal Bleeding. Can J Gastroenterol Hepatol. 2018 Jul 10;2018:3015891. doi: 10.1155/2018/3015891. eCollection 2018. PMID 30079329